CLINICAL TRIAL: NCT01141764
Title: Cerebral Metabolic Changes Associated With Thalamic Stimulation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Very slow and infrequent recruitment, availability of the imaging procedure at Adult Centre
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Elysa Widjaja, Staff Neuroradiologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000014496
Record Dates: First submitted 2010-06-07; First posted 2010-06-10 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Epilepsy
Keywords: pediatrics; Epilepsy; Deep Brain Stimulation; Positron Emission Tomography
MeSH Terms: conditions — Epilepsy | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): In our study, patients will be scanned with their DBS electrodes turned "on" and "off".
  Participation involves undergoing 2 separate PET scans on 2 separate days. The MRI and neuropsychological tests will either be performed on the same day as one of the PET scans or on a separate day.
  Procedures performed in this study are not part of the standard management of epilepsy.
  Interventions: Procedure: Positron Emission Tomography (PET) Scan; Procedure: Magnetic Resonance Imaging (MRI); Other: Neuropsychological Testing

INTERVENTIONS:
Procedure: Positron Emission Tomography (PET) Scan — The PET procedure consists of an intravenous injection of 18F-FDG followed by a 45-minute period of quiet resting. PET images will be acquired on an integrated PET/CT scanner.
  This process will be repeated with the stimulator "on" during the first PET image acquisition and "off" during the second PET image acquisition. "On" and "off" PET image acquisitions will be performed on two separate days.
Procedure: Magnetic Resonance Imaging (MRI) — MRI will be performed on a 1.5T system, using a combination of different sequences including sagittal T1, coronal and axial T2, FLAIR and proton density and axial 3D T1 weighted images.
Other: Neuropsychological Testing — On the same day or separate visit, depending on the timing of the PET imaging, they will be required to attend one half-day session for neuropsychological testing. Patients will arrive at the Toronto Western Hospital, the stimulator will be turned "off" for 30 minutes prior to neuropsychological testing with testing repeated with the stimulator on.

SUMMARY:
The purpose of this research study is to evaluate the brain circuits function and circuits involved in the mechanism of thalamic DBS in patients with medically refractory epilepsy.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) of the anterior nucleus of the thalamus in patients with medically refractory epilepsy has been shown to be efficacious. Studies have estimated a 46-76% reduction in seizures relative to the baseline. However, the exact anatomic circuitry involved in the mechanism of DBS in epilepsy remains unknown. Positron emission tomography (PET) studies can provide clues to the metabolic activity associated with DBS activation. In our study, patients will be scanned with their DBS electrodes turned "on" and "off". PET data captured during these two distinct states may show characteristic differences in cerebral glucose metabolism and modulatory effects of surrounding cerebral structures, thus providing clues to how DBS works to prevent seizures.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old
* currently have DBS implanted for medically refractory epilepsy
* Women of childbearing age will be required to use established contraceptive methods while enrolled in the study.

Exclusion Criteria:

Patients who:

* are < 18 years of age or > 85 years of age
* are medically unstable
* are women who are potentially pregnant, pregnant or nursing
* have had PET imaging within 1 year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Areas of the brain with low activity | within 30 days of enrollment in the study
  This measure will be based on the results of two PET scans done on separate days. The stimulator will be "on" during the first PET image acquisition and "off" during the second PET image acquisition.

SECONDARY OUTCOMES:
Brain Abnormalities | within 30 days of enrollment in the study
  One Magnetic Resonance Imaging (MRI) scan will be used to take detailed images of the brain and detect whether there are any abnormalities.
Ability to learn and understand | within 30 days of enrollment in the study
  One session of neuropsychological testing will be done in order to assess the subject's ability to learn and understand.

CONTACTS AND LOCATIONS:
Overall Officials: Elysa Widjaja, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (2):
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario